CLINICAL TRIAL: NCT01482416
Title: Flow-mediated Evaluation of the Brachial Artery of Climacteric Women Using Estradiol and Placebo. Randomized, Double Blinded, Placebo Controlled Study.
Brief Title: Vascular Effect of Estrogens Versus Placebo Evaluated by Flow-mediated Dilatation of Brachial Artery
Acronym: EDILA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Selmo Geber, Associate Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E.FR - 245365
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Unspecified Injury of Brachial Artery, Left Side, Initial Encounter
Keywords: hormone replacement therapy; Doppler velocimetry; Flow-mediated dilation; menopause
MeSH Terms: interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estrogen use (Experimental): climacteric women will use conjugated equine estrogens
  Interventions: Drug: Estrogens, Conjugated (USP)
- use of Placebo (Placebo Comparator): climacteric women will use placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estrogens, Conjugated (USP) — Experimental group will use 0.625mg/day during 30 days
  Other Names: Premarin
  Arms: Estrogen use
Drug: Placebo — Placebo group will use placebo once/day during 30 days
  Arms: use of Placebo

SUMMARY:
The aim of this study is to evaluate the vascular effects of estrogens on climacteric women measured by flow-mediated evaluation of the brachial artery using high resolution ultrasound and compare to placebo.

DETAILED DESCRIPTION:
The interruption of the secretion of sex steroids that occurs after menopause, determines a change in vascular pattern at various levels. As a result, several side effects might appear and interfere with women's quality of life and health. The use of hormone replacement therapy has contributed to the improvement in these effects. It has been observed vascular beneficial effects of sex steroids in premenopausal women, and of hormone replacement therapy (HRT) in climacteric women, on the central retinal arteries. The objective of this study is to evaluate the effects of conjugated equine estrogen on flow-mediated dilation of the brachial artery.

ELIGIBILITY:
Inclusion Criteria:

* Women without menstrual cycles within the last 12 months and FSH > 30IU/L
* Healthy women
* Women that were not using drugs with potential vascular effect within the last 1 year
* Women that never used hormone replacement therapy

Exclusion Criteria:

* Smoking
* Blood Pressure > 160/90 mm Hg.
* Breast and or endometrial cancer
* History of acute myocardial infarction
* Diabetes
* Vaginal bleeding of any origin
* Hepatic disease
* Thrombophlebitis or thromboembolic disorders

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the brachial artery | one month after treatment started
  Flow-mediated dilation will be measured by high resolution ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Selmo Geber, MD PhD, Principal Investigator — Medical School of Universidade Federal de Minas Gerais
Locations (1):
- Hospital das Clinicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Faria AF, de Souza MA, Geber S. Vascular resistance of central retinal artery is reduced in postmenopausal women after use of estrogen. Menopause. 2011 Aug;18(8):869-72. doi: 10.1097/gme.0b013e31820cc60c. PMID 21471823
- [Derived] Hurtado R, Celani M, Geber S. Effect of short-term estrogen therapy on endothelial function: a double-blinded, randomized, controlled trial. Climacteric. 2016 Oct;19(5):448-51. doi: 10.1080/13697137.2016.1201809. Epub 2016 Jul 16. PMID 27427235